CLINICAL TRIAL: NCT00002374
Title: A Phase IIIB Open-Label Trial Replacing Saquinavir HGC (Ro 31-8959) With Saquinavir SGC (Ro 31-8959) in Combination With Other Antiretroviral Drugs in Patients With HIV-1 Infection
Brief Title: A Study of Saquinavir Soft Gelatin Capsules Combined With Other Anti-HIV Drugs in HIV-1 Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229G; NR15521
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; HIV Protease Inhibitors; RNA, Viral; Saquinavir; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ritonavir; Nelfinavir; Saquinavir; Stavudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Saquinavir
Drug: Stavudine

SUMMARY:
To examine the efficacy of saquinavir SGC (soft gel capsules) in combination with other antiretrovirals in HIV-1 infected patients currently treated with saquinavir HGC (hard gel capsules) measured by the absolute change in plasma HIV-1 RNA during the 24 weeks of study treatment.

DETAILED DESCRIPTION:
Eligible patients will be stratified by HIV-1 RNA level into 2 populations: 1) >= 5,000-30,000 HIV-1 RNA, 2) > 30,000 HIV-1 RNA. All patients will be randomized to 1 of 3 treatment arms: Arm A - Saquinavir soft gel capsules (SQV SGC) + 2 new nucleoside analogs (reverse transcriptase inhibitors [RTIs]), Arm B - SQV SGC + nelfinavir + stavudine (d4T) or a new RTI, or Arm C - SQV SGC + ritonavir + d4T or a new RTI. All patients will undergo plasma HIV-1 RNA determinations, CD4 lymphocyte counts, hematology and chemistry blood work at baseline, weeks 4, 8, 12, 16 and 24.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 > 100 cells/mm3.
* Saquinavir HGC-experienced patients (>= 3 months cumulative therapy).

Required:

>= 3 months cumulative saquinavir HGC therapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Pacific Oaks Med Ctr, Beverly Hills, California
  - Tower Infectious Diseases / Med Associates Inc, Los Angeles, California
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - Ctr for Quality Care, Tampa, Florida
  - Community Research Initiative of New England, Brookline, Massachusetts
  - AIDS Ctr, New York, New York
  - Anderson Clinical Research / Inc, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Cadman J. Roche brings new formulation of saquinavir to FDA. Food and Drug Administration. GMHC Treat Issues. 1997 Apr-May;11(4/5):8. PMID 11364377